CLINICAL TRIAL: NCT02482259
Title: Assessment of Frailty in Patients With Advanced Hepatocellular Cancers
Acronym: FAC-L
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 6730
Record Dates: First submitted 2015-06-12; First posted 2015-06-26 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Hepatocellular Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is looking at the feasibility of performing frailty assessments on patients with advanced hepatocellular cancer.

DETAILED DESCRIPTION:
This study is primarily looking to see if it is feasible to assess frailty in patients with advanced hepatocellular cancer. It is also evaluating whether there may be any correlation between these assessments and toxicity of treatment and outcome.

The assessments include: Frailty score, nutritional assessment, comorbidity score and quality of life. In addition sarcopenia will be assessed measuring muscle mass from imaging performed as part of routine clinical care.

The assessments will be performed at baseline on entry into the study, at week 9 and week 18.

There is the option for patients to also donate a blood samples for research purposes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of hepatocellular cancer not suitable for curative treatment
* Seen by an oncologist or hepatologist for consideration of palliative treatment and a decision regarding management already made
* WHO Performance status 0-2
* Childs Pugh Score A or B
* Written informed consent

Exclusion Criteria:

N/A

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Hepatocellular cancer
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2016-07-19 (Actual); Study Completion 2016-07-19 (Actual)

PRIMARY OUTCOMES:
Percentage patients consenting for assessment out of number of patients approached | baseline
  Number of patients consenting for the study as a percentage of the number of patients approached about the study
Time taken to complete assessments | Baseline, week 9 and week 18
  Time taken to completed assessments recorded by clinical trials officer

SECONDARY OUTCOMES:
Frailty as a predictor of grade 3/4 toxicity | Baseline, week 9 and week 18
  Frailty score at baseline and during study time predict for outcome
Muscle mass and timed get up and go as predictors of outcome | Baseline, week 9 and week 18
  muscle mass as measured on routine CT scans and get up and go as measured in frailty score

OTHER OUTCOMES:
Quality of Life - EORTC QCQ 30 and HCC18 | Baseline, week 9 and week 18
Biomarker assessment of frailty and associated factors | Baseline, week 9 and week 18

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Plummer, MD, MRCP, BA, DPhil, Principal Investigator — Newcastle Unversity
Locations (1):
- Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, United Kingdom